CLINICAL TRIAL: NCT06184997
Title: Effect of a Sugar-free Isotonic Drink on Different Health Bioparameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, Prof. Dr. Alejandro Martínez-Rodríguez, Full professor, University of Alicante
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UA-2023-10-03
Record Dates: First submitted 2023-12-14; First posted 2023-12-29 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to group A (water, placebo) or group B (sugar-free isotonic drink), and will be instructed to consume 265 ml of water or 265 ml of sugar-free isotonic drink, respectively, every day for 12 weeks. During the study period, participants will be advised to maintain their usual diet and physical activity.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be aware that there are other people consuming a different type of drink than theirs. The person analyzing the results will also be unaware. However, the researchers will be aware because they need to control the supply.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (Placebo Comparator): Volunteer participants who will drink water
  Interventions: Other: PLACEBO
- ISOTONIC DRINK GROUP (Experimental): Volunteer participants who will drink Natural isotonic drink based on 20% Atlantic sea water, mixed with lemon and stevia.
  Interventions: Other: INTAKE OF ISOTONIC DRINK

INTERVENTIONS:
Other: INTAKE OF ISOTONIC DRINK — Intake of natural isotonic drink based on 20% Atlantic sea water, mixed with lemon and stevia.
  Arms: ISOTONIC DRINK GROUP
Other: PLACEBO — Intake of natural mineral water
  Arms: CONTROL GROUP

SUMMARY:
Randomized clinical trial in which 160 participants (80 men, 80 women) will be assigned to one of two groups (40 participants per group), to determine the effects of isotonic drink on different health parameters, following published recommendations. Subjects will be electronically randomized by block design into two arms: an experimental group: isotonic drink and a control group (placebo): normal water.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged >18 years;
* body mass index (BMI) of 18 to 25 kg/m^2;

Exclusion Criteria:

* individuals who have taken medication up to 3 months before the start of the study or supplements during the study;
* individuals with a history of gastrointestinal pathology or disorder such as duodenal ulcer, chronic colitis, or chronic inflammatory disease/surgery of the gastrointestinal tract (Crohn's disease, ulcerative colitis), celiac disease, or irritable bowel syndrome;
* individuals with serious acute or chronic diseases, treatments, or recent surgery;
* individuals with a report of serum levels of aspartate aminotransferase (AST), alanine aminotransferase (ALT), or gamma-glutamyl transferase (GGT) above the upper limit of the reference interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Body composition | 12 weeks
  Measurement of body composition using bioimpedance with the Biodyxpert device.
Body composition | 12 weeks
  Measurement of body composition through anthropometry.
Blood pressure | 12 weeks
  Measurement of systolic and diastolic blood pressure. Using an OMROM upper arm blood pressure monitor.
Perception of quality of life | 12 weeks
  Using a Quality of Life Questionnaire (SF36). Quality of Life Questionnaire is a comprehensive questionnaire that covers various attributes of an individuals life. It covers a variety of demographic questions to get better quality data and information before analyzing the quality of life of an individual.The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Perceived stress | 12 weeks
  Measurement of perceived stress using the Perceived Stress Scale (PSS)
BLOOD GLUCOSE | 12 weeks
  Glucose levels in blood by blood analysis.
BLOOD INSULIN | 12 weeks
  Insulin levels in blood by blood analysis.
BLOOD LIPID PORFILE | 12 weeks
  Cholesterol and triglycerides levels in blood.
Specific color of urine | 12 weeks
Specific gravity of urine | 12 weeks
Minerals in urine | 12 weeks
  K+ (Potassium), Na+ (Sodium), Mg2+ (Magnesium), Ca2+ (Calcium)
Urinary pH | 12 weeks
Mood States Profile | 12 weeks
  The POMS (Profile of Mood States) questionnaire is a psychological assessment tool widely used to measure mood states. It consists of a series of words or phrases that describe feelings and emotions. Participants are asked to rate each item on a scale, indicating how well it represents their mood over a specific period. The POMS measures six different mood dimensions: Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. It's commonly used in clinical settings, as well as in research studies, to assess the impact of various treatments or interventions on mood states. The POMS is valued for its sensitivity in detecting mood changes over time and its ability to differentiate between various mood states.
Evaluation of constipation symptoms by the patient | 12 weeks
  The PAC-SYM (Patient Assessment of Constipation Symptoms) is a self-report questionnaire designed to evaluate the symptoms of constipation from the patient's perspective. It is commonly used in clinical research and practice to assess the severity and impact of constipation symptoms. The questionnaire includes a series of items that ask patients to rate the frequency and severity of their constipation-related symptoms, such as abdominal discomfort, straining, and incomplete bowel movements.
Evaluation of the quality of life of patients with constipation (PAC-QOL) | 12 weeks
  The PAC-QOL (Patient Assessment of Constipation Quality of Life) questionnaire is a specialized tool designed to assess the quality of life in individuals suffering from constipation. It is a patient-reported outcome measure that focuses on how constipation affects a person's daily life, well-being, and overall health.
Sleep quality | 12 weeks
  Measurement of sleep quality using the Pittsburgh sleep quality index.
Liver biomarkers | 12 weeks
  Measurement of liver biomarkers through a blood test; Aspartate aminotransferase (AST or GOT), Alanine aminotransferase (ALT or GPT) and Bilirubin
Microbiome Indices | 12 weeks
  Microbiome indices through stool sample; Firmicutes/Bacteroidetes, Bacteroides/Prevotella, Enterobacteria/Enterococcus, Clostridium coccoides/perfringens

SECONDARY OUTCOMES:
Weight | 12 weeks
  Weight evaluation using a digital scale

CONTACTS AND LOCATIONS:
Locations (1):
- Alejandro Martínez Rodríguez, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No